CLINICAL TRIAL: NCT06519188
Title: The Effect of Salt Water Application on Cough, Sputum, Dyspnea Management and Quality of Life in Individuals With Chronic Obstructive Pulmonary Disease
Brief Title: The Effect of Salt Water Nebulization on Cough, Sputum and Quality of Life in Chronic Obstructive Pulmonary Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Turkey (Other Government)
Responsible Party: Principal Investigator, Zeliha Ermiş, Head Investigator, Ministry of Health, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Salt Water Nebulization
Record Dates: First submitted 2024-06-30; First posted 2024-07-25 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Copd
Keywords: quality of life; cough; dyspnea; COPD; saline water; nursing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cough; Dyspnea | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: pretest, posttest randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEBUL APPLICATION GROUP (Experimental): The experimental group patients were taught the method of nebulization with 5 ml isotonic sodium chloride. Patients were asked to perform the application twice a day, in the morning and in the evening, for two months.
  Interventions: Other: Nebulization application with 5 ml isotonic sodium chloride
- NON APLICATION GROUP (No Intervention): No intervention was performed on control group patients who volunteered for the study.

INTERVENTIONS:
Other: Nebulization application with 5 ml isotonic sodium chloride — Nebulization application with 5 ml isotonic sodium chloride in the morning and evening for two months.
  Arms: NEBUL APPLICATION GROUP

SUMMARY:
The aim of this clinical trial is to evaluate the effects of salt-water nebulization on individuals with chronic obstructive pulmonary disease. The main questions it aims to answer are:

Does salt-water application have an effect on cough and sputum management in individuals with COPD diagnosis? Does salt-water application have an effect on dyspnea management in individuals with COPD diagnosis? Does salt-water application have an effect on the quality of life in individuals with COPD diagnosis? The work was continued with two groups that did and did not practice. The group who made the application made the application twice a day every day for 2 months. The results of both groups were compared.

DETAILED DESCRIPTION:
In order to ensure randomization, the control group patient was selected on one day of the week and on the other day of the experiment. The patients were selected to be 50 people in the experimental group and 50 people in the control group. The experimental group was completed with 37 patients and the control group with 44 patients. The data were collected from the Patient Information Form, Modified Medical Research Council Scale/Medical Research Board Scale (MMRC), COPD Assessment Test (CAT), St. George was collected by Respiratory Survey. SPSS (IBM SPSS Statistics 27) package program was used for statistical analysis. Descriptive statistics and frequency tables were used in the interpretation of the findings. Parametric methods were used for the measurement values in accordance with the normal distribution. In accordance with parametric methods, the "Paired-Sample" test (t-table value) method was used to compare the measurement values of the two dependent groups. Non-parametric methods were used for measurement values that do not correspond to the normal distribution. In accordance with non-parametric methods, the "Mann-Whitney U" test (Z-table value) was used to compare the measurement values of two independent groups, and the "Friedman" test (χ2-table value) was used to compare the measurement values of three or more dependent groups. The "Pearson-χ2" cross tables were used to examine the relationships of the two qualitative variables to each other. The "Spearman" correlation coefficient was used to examine the relationships of two quantitative variables with each other.

ELIGIBILITY:
Inclusion Criteria:

* 35 years and above,
* Volunteer to participate in the research,
* Diagnosed with Stable COPD by the physician,
* Those who have not had an attack in the last month (are stable in terms of drug treatment),
* Having no vision, speech or hearing problems that would prevent understanding and applying the information given,
* Those who have smoked for at least 10 years or more,
* Individuals who are mentally competent (without intellectual disability).

Exclusion Criteria:

* Those who do not want to participate in the research,
* Hearing-speech impaired,
* Unable to communicate due to speaking different languages,
* Patients diagnosed by a physician with hypertension, ischemic heart disease, congestive heart failure, atrial fibrillation, chronic renal failure, stroke and other cerebrovascular disease, angina, major psychiatric disease (dementia, schizophrenia, etc.).

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The effect of salt water application on cough in individuals diagnosed with COPD after a 8 weeks period. | Base week and measurement interval is 8 weeks.
  COPD Assesment Test's 1st question is belong to cough. The cough assessment of the patients was evaluated from "0" (no cough) to "5" (a lot of coughing). As the score obtained from the scale increases, the rate of being affected by COPD also increases.
The effect of salt water application on sputum management in individuals diagnosed with COPD after a 8 weeks period. | Base week and measurement interval is 8 weeks.
  COPD Assesment Test's 2nd question is belong to sputum. The sputum assessment of the patients was evaluated from "0" (no sputum) to "5" (a lot of sputum). As the score obtained from the scale increases, the rate of being affected by COPD also increases.

SECONDARY OUTCOMES:
The effect of salt water application on dyspnea management in individuals diagnosed with COPD after a 8 weeks period. | Base week and measurement interval is 8 weeks.
  The Modified Medical Research Council Scale dyspnea scale is a five-item scale based on various physical activities that create a feeling of dyspnea.
  In this scale, "0" (NO DYSPNEA) and "4" (WORST DYSPNEA). As the score obtained from the scale increases, the rate of being affected by COPD also increases.
The effect of salt water application on quality of life in individuals diagnosed with COPD after a 8 weeks period. | Base week and measurement interval is 8 weeks.
  St. George's Respiratory Questionnaire with Quality of life were monitored in patients every 14 days and for the following 8 weeks.
  A score of zero (0) Good state of health, and (100) indicates the most severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: ZELIHA ERMIS, Principal Investigator — MOH TURKEY
Locations (1):
- Yedikule Chest Surgeory and Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The part of this study that can be shared is the statistical information and results.